CLINICAL TRIAL: NCT03300063
Title: Effects of Treating Sleep Apnea-Induced Hypoxemia With Low-Flow Oxygen in Acute Stroke Patients: A Pilot Study
Brief Title: Treating Sleep Apnea Induced Hypoxemia With Oxygen in Acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Melissa Lipford, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-002975
Record Dates: First submitted 2017-08-28; First posted 2017-10-03 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Standard Medical care
- Low Flow Nocturnal Oxygen (Active Comparator): This group will receive standard medical care as well as low flow oxygen during sleep.
  Interventions: Other: Low flow nocturnal oxygen

INTERVENTIONS:
Other: Low flow nocturnal oxygen — Nocturnal low-flow oxygen via nasal cannula
  Arms: Low Flow Nocturnal Oxygen

SUMMARY:
We want to determine if treating acute ischemic stroke patients who have evidence of hypoxemia due to sleep apnea with low flow O2 during sleep might help improve clinical and functional outcomes.

DETAILED DESCRIPTION:
Acute stroke patients will be tested for nocturnal hypoxemia using overnight oximetry. Those with evidence of hypoxemia will be randomized into two groups. One group will receive standard medical care. The other group will receive standard medical care as well as receiving low flow oxygen during sleep.

ELIGIBILITY:
Patients presenting to Mayo Clinic Hospital with acute ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Melissa C Lipford, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials